CLINICAL TRIAL: NCT00112528
Title: Phase II Trial of Bevacizumab, Gemcitabine, Oxaliplatin in Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Bevacizumab, Gemcitabine, and Oxaliplatin in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N034A; NCI-2012-02655 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000430845 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatic Cancer
Keywords: duct cell adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine + bevacizumab + oxaliplatin (Experimental): Patients receive gemcitabine IV over 100 minutes and bevacizumab IV over 30-90 minutes on days 1 and 15. Patients also receive oxaliplatin IV over 120 minutes on days 2 and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 courses of therapy beyond CR.
  After completion of study treatment, patients are followed every 3-6 months for up to 5 years.
  Interventions: Biological: bevacizumab; Drug: gemcitabine hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with gemcitabine and oxaliplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with gemcitabine and oxaliplatin works in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 6-month survival of patients with metastatic adenocarcinoma of the pancreas treated with bevacizumab, gemcitabine, and oxaliplatin.

Secondary

* Determine the objective response rate in patients with measurable disease treated with this regimen.
* Determine median survival, progression-free survival, time to treatment failure, and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 100 minutes and bevacizumab IV over 30-90 minutes on days 1 and 15. Patients also receive oxaliplatin IV over 120 minutes on days 2 and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 courses of therapy beyond CR.

After completion of study treatment, patients are followed every 3-6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed ductal cell or undifferentiated adenocarcinoma of the pancreas

  * Previously untreated metastatic disease
* No islet cell or acinar cell carcinoma or cystadenocarcinoma
* No invasion of adjacent organs (i.e., duodenum or stomach) or major blood vessels ( i.e., superior mesenteric artery or celiac artery)
* No CNS metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* No bleeding diathesis or uncontrolled coagulopathy
* No bleeding events within the past 6 months

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN) (stenting allowed)
* AST ≤ 5 times ULN
* No esophageal varices

Renal

* Creatinine ≤ 2 times ULN
* Proteinuria < 1+ by dipstick or urinalysis OR
* Protein < 1 g/24-hr urine collection
* No nephrotic syndrome

Cardiovascular

* No New York Heart Association class II-IV congestive heart failure
* No symptomatic, unstable angina, or coronary artery disease
* No uncontrolled cardiac arrhythmias
* No myocardial infarction within the past 6 months
* No uncontrolled hypertension
* No history of cerebrovascular events
* No clinically significant peripheral arterial disease
* No other clinically significant cardiac disease

Pulmonary

* No hemoptysis within the past 6 months

Immunologic

* No history of allergy or hypersensitivity to bevacizumab, oxaliplatin, or gemcitabine
* No hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No known allergy to other platinum compounds
* No ongoing or active infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No serious, non-healing wound, ulcer, or bone fracture
* No pre-existing peripheral neuropathy > grade 1
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or prostate cancer with a Gleason score < 7
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No gastrointestinal bleeding within the past 6 months
* No unresolved physical trauma within the past 4 weeks

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 months since prior immunotherapy or biologic therapy
* No prior adjuvant bevacizumab
* No concurrent immunotherapy
* No concurrent colony-stimulating factors during the first course of study therapy

Chemotherapy

* Recovered from prior chemotherapy
* More than 4 months since prior adjuvant chemotherapy for completely resected disease
* At least 4 months since prior chemoradiotherapy for locally advanced disease
* More than 4 months since prior gemcitabine as a radiosensitizer or as maintenance therapy
* No prior cytotoxic chemotherapy for metastatic disease
* No prior adjuvant oxaliplatin
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* More than 4 months since prior radiotherapy
* No prior radiotherapy to > 25% of bone marrow
* No prior radiotherapy to sole site of measurable disease unless there is radiologically confirmed progression of the irradiated tumor
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery or trauma and recovered
* No concurrent surgery

Other

* More than 2 weeks since prior and no concurrent thrombolytic agents

  * Anticoagulation therapy with warfarin or low molecular weight heparin is allowed provided the following criteria are met:

    * At least 2 weeks at a stable dose
    * INR 2-3
    * No active bleeding or pathologic condition that confers a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* No recent or concurrent participation in another study of experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-06; Primary Completion 2006-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Survival at 6 months | at 6 months

SECONDARY OUTCOMES:
Objective response rate as measured by RECIST criteria | Up to 5 years
Median survival | Up to 5 years
Progression-free survival | Up to 5 years
Time to treatment failure | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: George P. Kim, MD, Study Chair — Mayo Clinic
Locations (201):
- United States (201):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thorton, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, P. C., Ames, Iowa
  - Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Ottumwa Regional Health Center Cancer Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Sartell, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Bryan LGH Medical Center - West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Kim GP, Alberts SR, Oberg AL, et al.: Phase II trial of bevacizumab, gemcitabine, and oxaliplatin in patients with metastatic pancreatic adenocarcinoma. [Abstract] American Society of Clinical Oncology 2007 Gastrointestinal Cancers Symposium, 19 -21 January 2007, Orlando, Florida A-169, 2007.